CLINICAL TRIAL: NCT05023772
Title: A Clinical Trial Evaluating the Efficacy of Combining Laser Interstitial Thermal Ablation With and Without Spine Stereotactic Radiosurgery for Patients With Spine Metastases
Brief Title: Laser Interstitial Thermal Ablation and Stereotactic Radiosurgery for Patients With Spine Metastases
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Ian Lee, MD, Co-Director of the Hermelin Brain Tumor Center, Henry Ford Health System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14622
Record Dates: First submitted 2021-07-02; First posted 2021-08-27 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Neoplasm Metastasis; Spinal Cord Diseases; Spinal Cord Compression; Spinal Cord Tumor; Spine Metastases
Keywords: Laser Ablation; Spinal Cord; Minimally Invasive Surgical Procedure; Stereotactic Radiosurgery; Pain Control; Metastasis; Epidural Tumor
MeSH Terms: conditions — Neoplasm Metastasis; Spinal Cord Diseases; Spinal Cord Compression; Spinal Cord Neoplasms; Agnosia; Epidural Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Intervention Model Description: Open Label one arm. Unblinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Experimental Treatment of Laser Interstitial Thermal Ablation Therapy and Stereotactic Radiosurgery (Experimental): Patients will undergo laser interstitial thermal ablation and CT guided stereotactic radiosurgery via intensity-modulated radiation therapy on different dates within a one to fourteen day window. The order of treatment is at the treating physicians discretion.
  Interventions: Procedure: Stereotactic Laser Ablation; Radiation: Stereotactic Radiosurgery; Diagnostic Test: MRI guided laser ablation

INTERVENTIONS:
Procedure: Stereotactic Laser Ablation — MR Guided laser ablation therapy
  Other Names: Thermal laser ablation therapy; Visualase laser ablation therapy
Radiation: Stereotactic Radiosurgery — Precise delivery of radiation to spinal tumor
  Other Names: CT guided stereotactic radiosurgery; Stereotactic external beam radiation therapy
Diagnostic Test: MRI guided laser ablation — Surgery will take place in intraoperative suite to include operating room and MRI scanner
  Other Names: Intraoperative MRI

SUMMARY:
The purpose of this research is to combine two complementary modes of treatment, spinal interstitial laser ablation and stereotactic spine radiosurgery (SSRS) for the treatment for spinal tumors near the spinal cord with an objective to improve tumor control, improve pain control, preserve function, and improve quality of life. We will also assess how effective these combined modes of treatment are in patients with spinal metastasis with an epidural component.

DETAILED DESCRIPTION:
Primary Objectives:

1. Documenting rate of local control in patients who have received this combined treatment and
2. Documenting safety of MRI compatible hardware for MRI based image guidance
3. Determining the accuracy of the MRI-based image guidance

Secondary Objectives:

1. To determine local control at 1, 3, 6, 9, 18, and 24 months, and to compare to a historical control where patients received only SSRS at these time points and at 12 months.
2. To document the extent of epidural tumor regression at 1, 3, 6, 9, 12, 18 and 24 months

   * Calculate decrease in epidural tumor volume (by volumetric measurements using Brain Lab Elements software)
   * Calculate increase in thecal sac patency (by volumetric measurements using Brain Lab Elements software and according to Bilsky method
3. To determine overall survival at 6, 12, 18, and 24 months.
4. To assess changes in muscle strength, location and severity of spinal-related pain, sensory function, ability to ambulate, and neurological grading at 1, 3, 6, 9, 12, 18, and 24 months compared with pretreatment baselines.
5. To assess the effect of treatment on quality of life, measured at 1 month and every 3 months after with validated outcome measure tools
6. To describe adverse side effects after treatment and to descriptively correlate those effects with radiographic findings, pain control, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old. (The indication for this technique is controversial in skeletally immature patients.)
* Histologic diagnosis of solid malignant tumor (not one of the more radiosensitive histologic subtypes, see Exclusion Criteria), including but not limited to non-small cell lung cancer, breast, prostate, renal cell, melanoma, gastrointestinal, sarcoma, thyroid, head and neck primary, and unknown primary tumors.
* Quantification of the degree of epidural spinal cord compression as grade 1C, 2, or 3 by MRI, with and without contrast sequences. Axial T2 sequence is encouraged but not required.
* The vertebral body site to be treated must be located from T2 to L1
* No more than 3 contiguous or dis-contiguous vertebral levels involved with metastasis in the spine to be irradiated in a single session or 3 sessions.
* Motor strength ≥4 out of 5 in extremity or extremities affected by the level of the spinal cord compression (see section 4 for grading method).
* ECOG performance status <2 or Karnofsky performance status (KPS) >50
* Life expectancy >3 months.
* Inoperable disease because of patient refusal, neurosurgical evaluation, or any other medical reasons.
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) before study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Prior conventional radiation to the same site is allowed as long as there is a greater than 3 months interval.
* Signed informed consent.

Exclusion Criteria:

* Requires open spinal procedure or a percutaneous procedure without the use of image guidance.
* Primary tumors of radiosensitive histology (lymphoma, multiple myeloma, small cell carcinoma, germ cell tumors), as conventional radiation is likely to be effective in such cases.
* Unable to tolerate general anesthesia and prone position.
* Unable to undergo MRI scan of the spine.
* Inability to lie flat on a treatment table for >60 minutes.
* Pregnant. (Urine testing must be done no more than 10 days prior to surgery.)
* Prior conventional irradiation of the spine site and level to be treated with an interval shorter than 3 months.
* Frank cord compression or cord compression from bone components or configuration and acute neurological deficits (defined as motor strength <4/5 in extremity or extremities affected by the level of the spinal cord compression)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-09-02 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12-20 (Estimated)

PRIMARY OUTCOMES:
Local Tumor Control Rate | up to 24 months
  Kaplan-Meier estimates will be used.

SECONDARY OUTCOMES:
Local Tumor Control | 1, 3, 6, 9, 12, 18, and 24 months
  Time to local failure will be monitored continuously using Bayesian method.
Postoperative response to treatment assessed by MRI | 1, 3, 6, 9, 12, 18, and 24 months
  Routine MRI of the spine with and without contrast will be obtained at each follow-up visit. These post-treatment scans will be analyzed and compared to baseline scans for assessment of treatment response and local control. Bilsky grading system will be used.
Adverse Events | up to 24 months
  To describe adverse side effects after treatment and descriptively correlate those effects with radiographic findings, pain control, and quality of life.
Overall Survival | 6, 12, 18, and 24 months
  Kaplan-Meier estimates will be used.
Changes in symptoms assessed by physical examination | 1, 3, 6, 9, 12, 18, 24 months and annually thereafter
  The Physical Exam includes a general exam:(HEENT) Head, Eye, Ear, Nose and Throat evaluation, chest, heart, abdomen and extremities exam. Changes will be compared to baseline measurements. Negative changes will be evaluated by the neurosurgeon and radiation oncologist to determine if the change is related to a local failure or progression of systemic disease. Kaplan-Meier estimates will be used.
Changes in symptoms assessed by neurological examination | 1, 3, 6, 9, 12, 18, and 24 months
  The neurological examination includes: mental status (tested through history taking), cranial nerves (observation of eyes, face, voice, and coordination during history taking and as patient moves about the exam room), motor system (visual inspection, tone, muscle strength and endurance, assigned score of 0-5 for each muscle, a score of 0 would mean no muscular contraction, and a score of 5 would mean movement against full resistance, normal strength), reflexes, sensory system (vibration in toes; pinprick in feet); coordination (truncal stability, fine finger movement, toe tapping, finger-nose-finger, heel-knee-shin), and station and gait (gait including arising from chair without hands, walking on toes, heels, and heel to toe). Kaplan-Meier estimates will be used.

OTHER OUTCOMES:
Measuring Quality of life (QOL) assessed by Spine Tumor Survey (MDASI-SP) | baseline and 1, 3, 6, 9, 12, 18, and 24 months
  We are measuring quality of life with the Spine Tumor Survey that will be assessed during each follow up Clinic visit. The patient survey will be assessed to measure postoperative response to treatment.
Measuring Quality of life (QOL) assessed by Health Survey (SF-36) | baseline and 1, 3, 6, 9, 12, 18, and 24 months
  We are measuring quality of life with the Health Survey that will be assessed during each follow up Clinic visit. The participants are asked questions that measure eight health domains to assess physical and mental health. Physical health-related domains include: General health, Physical Functioning, Role Physical, and Body Pain. Mental health-related scales include Vitality, Social Functioning, Role Emotional, and Mental Health. A 3 and 5 point Likert scale is used in the survey. Two summary scores of the physical and mental health using weighted means of the eight domains. Descriptive statistics will be used to summarize pain relief and quality of life at each follow up visit, which will be the changes in scores from baseline to each assessment visit. Time to maximum pain relief will be the time from the day of thermal ablation until the lowest pain score for average pain after radiotherapy.
Measuring Quality of life (QOL) assessed by Brief Pain Inventory Survey (BPI) | baseline and 1, 3, 6, 9, 12, 18, and 24 months
  We are measuring quality of life with the Brief Pain Inventory Survey that will be assessed during each follow up Clinic visit. The patient survey will be assessed to measure postoperative response to treatment. Participants are asked to assess the severity of pain and the impact of pain on daily functions. Severity of pain, including the pain location, worst pain in the last 24 hours, least pain in the last 24 hours, pain on average and pain right now. Range 0-10: a score of 0 would mean no pain and a score of 10 means the pain is as bad as you can imagine. Pain medications, amount of pain relief in the past 24 hours, and impact of pain on daily function, including general activity, mood, walking ability, normal work, relations with other people, sleep, enjoyment of life, and range 0-10.

CONTACTS AND LOCATIONS:
Overall Officials: Ian Lee, MD, Principal Investigator — Henry Ford Health Health System
Locations (1):
- Henry Ford Hospital, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-05-24): https://cdn.clinicaltrials.gov/large-docs/72/NCT05023772/ICF_001.pdf